CLINICAL TRIAL: NCT05160636
Title: Patient-Reported Outcomes Associated With COVID-19 and Influenza: A Prospective Survey Study on Outpatient Symptomatic Adults With Test-Confirmed Illness in the United States
Brief Title: A Study to Look at the Health Outcomes of Patients With COVID-19 and Influenza
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: CVS Caremark (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591034; NCT05160636 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-12-15; First posted 2021-12-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: COVID-19; Coronavirus Disease 2019; Influenza
Keywords: Patient-Reported Outcomes; Humanistic Burden; Quality of Life; Disease Symptoms Assessment; COVID-19; SARS-CoV-2; Severe Acute Respiratory Syndrome Coronavirus 2 Infection; Acute respiratory infection; Influenza; Human Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Nasopharyngeal swabs that are obtained as SOC for COVID-19 testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Positive: Test-confirmed COVID-19 illness and at least one patient-reported symptom
  Interventions: Biological: COVID-19 Vaccine
- Influenza Positive: Test-confirmed influenza illness and at least one patient-reported symptom

INTERVENTIONS:
Biological: COVID-19 Vaccine — Receipt of Pfizer BioNTech COVID-19 vaccine
  Groups: COVID-19 Positive

SUMMARY:
The main purpose of this study is to understand:

* the symptoms of COVID-19 or influenza- health-related outcomes of people with COVID-19 or influenza (influenza only included in updated study analyses)
* the potential effects of COVID-19 vaccines in people with COVID-19

This study will enroll participants who are:

* 18 years or older
* reported to have symptoms with tests that have confirmed illness. The tests can be taken at any of CVS pharmacy COVID-19 or influenza test sites.

The study will collect vaccine history information from participants who are ready to take part in the study. Participant will be emailed a form with questions about their health related to COVID-19 or influenza during multiple follow-ups over a 6-month period.

DETAILED DESCRIPTION:
This is a prospective non-interventional longitudinal cohort survey study. Repeated measures on PROs including: symptoms (prevalence, frequency, duration, and severity), EQ-5D-5L, and WPAI over 6 months will be collected and evaluated.

COVID-19 Cohort: Participants 18 years or older with test-confirmed COVID-19 illness and at least one patient-reported symptom.

Influenza Cohort: Participants 18 years or older with test-confirmed influenza illness and at least one patient-reported symptom.

All study objectives and outcomes will be assessed separately for the two study cohorts. Influenza cohort is only included in updated study analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-reported at least one symptom in the CVS Health pre-test screening questionnaire
* Positive result reported from diagnostic test for COVID-19 (or influenza in updated analysis)
* Evidence of a signed and dated informed consent through electronic consent process indicating that the participant has been informed of all pertinent aspects of the study
* Able to complete the questionnaires by themselves in English or Spanish

Exclusion Criteria:

- No symptoms reported in the study screening questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are 18 years or older who are self-reported symptomatic, who tested positive with RT-PCR at any of the approximately 5,000 CVSH COVID-test sites and consented to participate in the PRO study.
  Updated study analysis included participants 18 years or older who are self-reported symptomatic, with test-confirmed illness when tested at any of CVS pharmacy COVID-19 or influenza test sites, and consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life (HRQoL) using EQ-5D-5L | 6 months
  To assess the change in HRQoL using EQ-5D-5L before COVID-19 or influenza and over a 6-month period following the test-confirmed COVID-19 or influenza.
EQ-5D-5L Utility Index (UI) scores | 6 months
  To estimate the EQ-5D-5L UI scores and their change across six time points in a span of six months following the test-confirmed COVID-19 or influenza.
Visual Analog Scale (VAS) scores | 6 months
  To estimate the VAS scores and their change across six time points in a span of six months following the test-confirmed COVID-19 or influenza.
WPAI scores | 6 months
  To estimate the WPAI scores and their change across six time points in a span of six months following the test-confirmed COVID-19 or influenza.

SECONDARY OUTCOMES:
Prevalence and duration of SARS-CoV-2 symptoms | 6 months
  To characterize prevalence and duration of SARS-CoV-2 symptoms before COVID-19 and up to 6 months (acute phase and Long COVID).
Prevalence, Severity, and duration of influenza symptoms aggregated as index score area under the curve | 6 Months
  To characterize prevalence and duration of influenza symptoms before influenza and up to 6 months (acute phase and Long Flu). Outcome will be aggregated by assigning a point-scale to the symptom severity and calculating the area under the curve of the severity index score.
Fatigue before COVID-19 | 6 months
  To assess fatigue (using PROMIS questionnaire Fatigue short-form 8a) before COVID-19 and over a six-month follow-up.
Fatigue after COVID-19 | 6 months
  To estimate the PROMIS questionnaire Fatigue short-form 8a score and its change across six time points in a span of six months following the RT-PCR confirmed COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sun X, Di Fusco M, Lupton LL, Yehoshua A, Alvarez MB, Allen KE, Puzniak L, Lopez SMC, Cappelleri JC. Predictors of Long COVID Among Symptomatic US Adults Testing Positive for SARS-CoV-2 at a National Retail Pharmacy. Healthcare (Basel). 2024 Nov 21;12(23):2321. doi: 10.3390/healthcare12232321. PMID 39684943
- [Derived] Di Fusco M, Cappelleri JC, Yehoshua A, Craig KJT, Alvarez MB, Allen KE, Porter TM, Lopez SMC, Puzniak L, Sun X. Associations between symptom-based long COVID clusters and long-term quality of life, work and daily activities among individuals testing positive for SARS-CoV-2 at a national retail pharmacy. J Patient Rep Outcomes. 2024 Oct 22;8(1):122. doi: 10.1186/s41687-024-00797-7. PMID 39436613
- [Derived] Sun X, Di Fusco M, Puzniak L, Coetzer H, Zamparo JM, Tabak YP, Cappelleri JC. Assessment of retrospective collection of EQ-5D-5L in a US COVID-19 population. Health Qual Life Outcomes. 2023 Sep 8;21(1):103. doi: 10.1186/s12955-023-02187-x. PMID 37679771
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591034